CLINICAL TRIAL: NCT02128945
Title: Dosimetry and Biodistribution of [18F]-Fludarabine in Lymphoid Malignancies
Acronym: FLUDATEP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: CNRS, UMR ISTCT 6301, LDM-TEP Groupe, GIP Cyceron, Caen, France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-002796-18; 13-090
Record Dates: First submitted 2014-04-09; First posted 2014-05-01 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-01

CONDITIONS: Untreated B-Chronic Lymphocytic Leukemia or Diffuse Large B Cells Lymphoma Patients
Keywords: PET; Chronic lymphocytic Leukemia (CLL); Diffuse Large B Cells Lymphoma (DLBCL); Fludarabine
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FLUDATEP (Experimental): [18F] - Fludarabine PET/CT
  Interventions: Other: [18F] - Fludarabine PET/CT

INTERVENTIONS:
Other: [18F] - Fludarabine PET/CT — [18F] - Fludarabine PET/CT before treatment

SUMMARY:
The application of positron emission tomography with lymphoproliferative diseases today provides diagnostic and therapeutic information of major importance , especially in terms of speed and quality of response to treatment. The radiopharmaceutical used in clinical practice for this exam is fluorodeoxyglucose 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose ([18F]-FDG) . However , the uptake of this tracer is not elective in lymphoid tissues , with a lack of specificity. In addition , the avidity of this tracer is unequal according to the histological subtype (lack of sensitivity).

To try to improve the results of this clinical exploration of lymphoid malignancies, the investigators developed a new radiopharmaceutical ( [18F] - fludarabine ). The idea of transforming the fludarabine radiopharmaceutical is based on the existence of a fluorine atom in the molecule and the pharmacokinetic characteristics of this drug. The [18F]-Fludarabine is a new radiopharmaceutical reproducing the same dosage formulation of fludarabine , a drug used for the treatment of certain types of lymphoproliferative diseases, especially those where the tumor cells have a low proliferation kinetics . This drug is used in therapy in particular pharmacokinetic effect for a high affinity for the lymphoid tissue . Preclinical results on normal and lymphoma xenograft -bearing mice showed a specificity restricted to lymphoid tissue fixation with [18F]-Fludarabine compared with [18F]-FDG .

Based on these encouraging results , the investigators propose in this work to explore the Dosimetry and Biodistribution of [18F] - Fludarabine in human lymphoproliferative diseases : 1)A first group of patients with non-Hodgkin's large cell lymphomas in which it already has a wealth of experience in exploration [18F]-FDG, and 2) a second group of patients with chronic lymphocytic leukemia, where the results of the exploration [18F]-FDG are considered disappointing and did not, for this reason, experienced clinical development.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18
* Signed written informed consent
* Untreated stage B or C chronic lymphocytic leukemia
* Untreated diffuse large B-cell lymphoma
* Eligible for PET-CT
* The subject must be covered by a social security system

Exclusion Criteria:

* Age under 18
* Patients concurrently included in an investigational trial
* Weight over 120 kg
* pregnant women
* active infectious disease
* immune hemolytic anemia
* patients with creatinine clearance < 30 ml/mn
* corticosteroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Standardized measure of [18F]-Fludarabine uptake in tumor tissue. | Day 0 ([18F]-Fludarabine PET-CT day)
  Measure of the Standard Uptake Value (SUV) for each lesion.

SECONDARY OUTCOMES:
Calculation of the equivalent dose to all organs and evaluation of effective dose to the whole body | Day 0 ([18F]-Fludarabine PET-CT day)

OTHER OUTCOMES:
Distribution and temporal activity curve of [18F]-Fludarabine obtained for each organ and collection of possible adverse events. | Participants will be followed for a maximum of 9 days after [18F]-Fludarabine PET-CT.
  Collection of every adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain P CHANTEPIE, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- University Hospital, Caen, France